CLINICAL TRIAL: NCT02454959
Title: A Randomized, Phase III, Two-period, Open-label, Chronic-dosing (7 Days), Multicenter, Crossover Study to Assess the Efficacy, Safety and Pharmacokinetics of PT003 in Subjects With Moderate to Very Severe COPD With and Without a Valved Holding Chamber
Brief Title: Crossover Study to Assess the Efficacy of PT003 With and Without a Valved Holding Chamber in Subjects With Moderate to Severe COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PT003013
Record Dates: First submitted 2015-05-13; First posted 2015-05-27 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFF MDI (PT003) with Aerochamber (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI) with Aerochamber Plus Valved Holding Chamber
  Interventions: Device: GFF MDI (PT003) with Aerochamber
- GFF MDI (PT003) without Aerochamber (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI) without Aerochamber Plus Valved Holding Chamber
  Interventions: Device: GFF MDI (PT003) without Aerochamber

INTERVENTIONS:
Device: GFF MDI (PT003) with Aerochamber — Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI) with Aerochamber Plus Valved Holding Chamber
  Arms: GFF MDI (PT003) with Aerochamber
Device: GFF MDI (PT003) without Aerochamber — Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI) without Aerochamber Plus Valved Holding Chamber
  Arms: GFF MDI (PT003) without Aerochamber

SUMMARY:
This is a Randomized, Phase III, Two-period, Open-label, Chronic-dosing (7 Days), Multi-center, Crossover Study to Assess the Efficacy of PT003 in Subjects with Moderate to Severe COPD with and without a Valved Holding Chamber.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age and no older than 80 at Screening
* Women of non-child bearing potential or negative serum pregnancy test at Screening, and agrees to acceptable contraceptive methods used consistently and correctly Screening until 14 days after final visit.
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking
* Pre- and post-bronchodilator FEV1/FVC ratio of <0.70
* Post-bronchodilator FEV1 must be <80% predicted normal value, calculated using NHANES III reference equations, and the measured FEV1 must also be ≥30% of predicted normal value.

Exclusion Criteria:

* Significant diseases other than COPD, i.e., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study.
* Women who are pregnant or lactating or women of childbearing potential who are not using an acceptable method of contraception.
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma.
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Screening or during the Screening Period.
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Screening or during the Screening Period.
* Subjects who have clinically significant uncontrolled hypertension.
* Subjects who have cancer that has not been in complete remission for at least five years.
* Subjects with abnormal liver function tests defined as AST, ALT, or total bilirubin ≥1.5 times upper limit of normal at Screening and on repeat testing.
* Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated. Subjects with a diagnosis of open angle glaucoma who have intraocular pressure controlled with medication(s) are eligible.
* Subjects with symptomatic prostatic hypertrophy that is clinically significant in the opinion of the Investigator. Subjects with a trans-urethral resection of prostate (TURP) or full resection of the prostate within 6 months prior to Screening are excluded from the study.
* Subjects with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, Study Director — Pearl Therapeutics
Locations (6):
- United States (6):
  - Pearl Investigative Site, Clearwater, Florida
  - Pearl Investigative Site, Tampa, Florida
  - Pearl Investigative Site, Winter Park, Florida
  - Pearl Investigative Site, Charlotte, North Carolina
  - Pearl Investigative Site, Winston-Salem, North Carolina
  - Pearl Investigative Site, Gaffney, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, 2-period, open-label, chronic dosing (7 days), cross-over study conducted at 8 sites in the US.
Pre-assignment Details: Subject received one week of study treatment for each of the treatment periods, separated by a washout period of 7-14 days between treatments. Intent-to-treat (ITT) Population is used for Participant Flow. By-sequence tabulations of the data were not pre-specified.
Groups:
- Overall Study: All Randomized Patients
Period: Overall Study
Arm/Group | Overall Study
Started | 79
GFF MDI (PT003) With Aerochamber | 73
GFF MDI (PT003) Without Aerochamber | 77
Completed | 70
Not Completed | 9
Not completed — Protocol-Specified Criteria | 3
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2

BASELINE CHARACTERISTICS:
Population: The Modified-Intent-to-Treat (MITT) Population is a subset of the Intent-to-Treat (ITT) Population including subjects who received treatment and had post-treatment efficacy data for both treatment periods and is used for the baseline characteristics.
Groups:
- MITT Population: The Modified ITT (MITT) Population is a subset of the ITT Population including subjects who received treatment and had post dose efficacy data from both Treatment Periods. Data judged to be impacted by major protocol deviations were determined prior to unblinding and excluded. Statistical tabulations and analyses are by randomized treatment, but data obtained after subjects received an incorrect treatment have been excluded from the affected periods.
Arm/Group | MITT Population
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.5 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 34

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve for Change From Baseline in Forced Expiratory Volume in 1 Second (FEV1) From 0 to 12 Hours (AUC0-12) on Day 8
Description: AUC0-12 was calculated using the trapezoidal rule based on FEV1 assessments at pre-dose, and 15 minutes, 30 minutes, 1 hour, 2 hours, 4 hours, 8 hours, 10 hours, 11.5 hours, and 12 hours post-dosing of study drug. Primary Outcome was calculated using the trapezoidal rule and was modeled conditionally on baseline FEV1.
Time Frame: 7 days of treatment
Population: The primary analysis used the Modified-Intent-to-Treat (MITT) Population.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- GFF MDI (PT003) With Aerochamber: Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003 (GFF MDI) 14.4/9.6 µg BID with Aerochamber Plus Valved Holding Chamber
- GFF MDI (PT003) Without Aerochamber: Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003 (GFF MDI) 14.4/9.6 µg BID without Aerochamber Plus Valved Holding Chamber
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 67 | 68
Liter | 1.538 (0.0228) | 1.516 (0.0227)

2. Secondary Outcome: AUC0-12 on Day 8
Description: Pharmacokinetic Parameter AUC0-12 of Glycopyrronium by Treatment on Day 8
Time Frame: Day 8
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 56 | 56
h*pg/mL | 128.00 (85.63) | 111.39 (63.54)

3. Secondary Outcome: AUC0-12 on Day 8
Description: Pharmacokinetic Parameter AUC0-12 of Formoterol by Treatment on Day 8
Time Frame: Day 8
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 49 | 51
h*pg/mL | 75.46 (43.29) | 78.49 (39.17)

4. Secondary Outcome: Cmax on Day 8
Description: Pharmacokinetic Parameter Cmax of Glycopyrronium by Treatment on Day 8
Time Frame: Day 8
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 62 | 67
pg/mL | 34.03 (21.87) | 26.55 (15.11)

5. Secondary Outcome: Cmax on Day 8
Description: Pharmacokinetic Parameter Cmax of Formoterol by Treatment on Day 8
Time Frame: Day 8
Population: Pharmacokinetic Population
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 62 | 67
pg/mL | 12.53 (5.88) | 13.07 (7.50)

6. Secondary Outcome: Tmax on Day 8
Description: Pharmacokinetic Parameter tmax of Glycopyrronium by Treatment on Day 8
Time Frame: Day 8
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: h
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 62 | 67
h | 0.10 (21.87) [0.03 to 10.02] | 0.12 (15.11) [0.03 to 8]

7. Secondary Outcome: Tmax on Day 8
Description: Pharmacokinetic Parameter tmax of Formoterol by Treatment on Day 8
Time Frame: Day 8
Population: Pharmacokinetic Population
Measure: Median (Full Range); unit: h
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Number analyzed (Participants) | 62 | 67
h | 0.33 (21.87) [0 to 10.02] | 0.37 (15.11) [0.37 to 10.17]

ADVERSE EVENTS:
Time Frame: Adverse events collected from the time the subject signed consent up to the follow-up phone call 7-14 days after last dose of study drug.
Description: Any Adverse Events reported as starting during a Washout Period were assigned to the last randomized treatment received including those occurring during a Washout Period or the Follow-up Period. Serious adverse events collected from the time the subject signed consent up to 14 days following the last dose of study drug.
Arm/Group | GFF MDI (PT003) With Aerochamber | GFF MDI (PT003) Without Aerochamber
Serious Adverse Events (participants affected / at risk) | 1/74 | 2/78
Other Adverse Events (participants affected / at risk) | 3/74 | 8/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) With Aerochamber (N=74) | GFF MDI (PT003) Without Aerochamber (N=78)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI (PT003) With Aerochamber (N=74) | GFF MDI (PT003) Without Aerochamber (N=78)
Blood potassium increased (Investigations) | 0 (0) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vessel puncture site swelling (General disorders) | 1 (2) | 2 (4)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.